CLINICAL TRIAL: NCT04363554
Title: The Kidneys Ability to Concentrate and Dilute Urine in Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD) or Other Cause of Chronic Renal Disease Compared to Healthy Volunteers
Brief Title: The Kidneys Ability to Concentrate and Dilute Urine in Patients With Autosomal Dominant Polycystic Kidney Disease
Acronym: POVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Jesper Norgaard Bech, Head of University Clinic in Nephrology and Hypertension, Regional Hospital Holstebro
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: My-1-2017
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Polycystic Kidney, Autosomal Dominant; Chronic Kidney Diseases
Keywords: CYSTS; KIDNEYS
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Renal Insufficiency, Chronic; Cysts

STUDY DESIGN:
Intervention Model Description: A case control, randomized crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urine dilution test (Other): Urine dilution test
  Interventions: Other: Fluid intake
- Urine concentration test (Other): Urine concentration test
  Interventions: Other: Thirsting

INTERVENTIONS:
Other: Fluid intake — The participants will intake fluid
  Arms: Urine dilution test
Other: Thirsting — The participants will thirst
  Arms: Urine concentration test

SUMMARY:
The ability to concentrate and dilute urine is primarily regulated via vasopressin (AVP) dependent Aquaporin-2 water channels (AQP2 channels) in the kidney's collecting duct. Autosomal dominant polycystic kidney disease (ADPKD) is a common genetic disorder, characterized by the formation of cyst in the kidneys, causing gradual renal function-loss. Previous studies indicate that ADPKD patients have decreased urine concentration, higher plasma osmolality, and plasma AVP levels compared to healthy controls. Previous studies also indicate that ADPKD patients' dysregulated AVP is an important factor for the pathogenesis and progression of the disease. It is unclear whether ADPKD patients' ability to concentrate and dilute urine are different from those of other cause of chronic renal disease to the same degree. It is also unclear, what mechanisms cause the decreased ability to concentrate and dilute urine in chronic renal disease patients. The purpose of this trial is to investigate the difference in renal function during concentration and dilution test in a case-control, randomized, cross-examination study with ADKPD patients or other cause of chronic renal disease compared to healthy volunteers.

DETAILED DESCRIPTION:
The aim is to measure the difference in renal function, including kidney tubular function, blood pressure and vasoactive hormones in patients with Autosomal dominant polycystic kidney disease (ADPKD) or other chronic renal disease compared to healthy volunteers, during concentration and dilution test.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients: -age >18 years, diagnosis with ADPKD, informed consent, contraception for fertile women
* Patients with chronic kidney disease: age >18 years, diagnosis with chronic kidney disease other then ADPKD, informed consent, contraception for fertile women
* Healthy volunteers: age >18 years, healthy, informed consent, contraception for fertile women

Exclusion Criteria:

* ADPKD patients: Renal transplantation, operation in the kidney, Diabetes mellitus, neoplastic conditions, pregnancy, breastfeeding, unwillingness to participate, intolerance towards urine dilution or urine concentration test, alcohol or medical abuse, BP >170/110 despite regulation, unacceptable side effects to background medication (antihypertensive medicine) during the trial.
* Patients with chronic kidney disease: Renal transplantation, operation in the kidney, Diabetes mellitus, medullary cystic kidney disease, lithium nephropathy, neoplastic conditions, pregnancy, nursing, unwillingness to participate, intolerance towards urine dilution or urine concentration test, alcohol or medical abuse, BP >170/110 despite regulation, unacceptable side effects to background medication (antihypertensive medicine) during the trial.
* Healthy volunteers: Arterial hypertension, significant clinical signs of heart, lungs, liver, kidneys, endocrine, brain or neoplastic disorders, alcohol or drug abuse, medical treatment, smoking, pregnancy or breastfeeding, smoking, clinically significant abnormal findings in blood, urine tests or electrocardiogram, blood donation within the last month before the examination date in the first trial sequence, intolerance to or unacceptable side effects of urine concentration and urine dilution test

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

PRIMARY OUTCOMES:
free water clearance CH20 u-osm | 5 hours
  free water clearance (CH2O)
u-osm | 4 hours
  urine osmolality

SECONDARY OUTCOMES:
free water clearance | 5 hours
  free water clearance (CH2O)

CONTACTS AND LOCATIONS:
Overall Officials: My Malmberg, MD, Principal Investigator — Departments of medical research and medicine
Locations (1):
- Department of Medical Research, Regional Hospital Holstebro, Holstebro, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malmberg MH, Mose FH, Pedersen EB, Bech JN. Urine concentration ability is reduced to the same degree in adult dominant polycystic kidney disease compared with other chronic kidney diseases in the same CKD-stage and lower THAN in healthy control subjects - a CASE control study. BMC Nephrol. 2020 Aug 31;21(1):379. doi: 10.1186/s12882-020-02043-w. PMID 32867720